CLINICAL TRIAL: NCT03255954
Title: Interpersonal Counseling (IPC) for University Counseling Centers
Brief Title: IPC for University Counseling Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Amherst College (Unknown); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00119669
Record Dates: First submitted 2017-05-23; First posted 2017-08-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Interpersonal Counseling
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interpersonal Counseling-C (Experimental): Interpersonal Counseling for University Counseling Centers is a psychotherapeutic intervention
  Interventions: Other: Interpersonal Counseling for University Counseling Centers

INTERVENTIONS:
Other: Interpersonal Counseling for University Counseling Centers — Interpersonal Counseling (IPC) is a brief version of Interpersonal Psychotherapy (IPT). IPC synthesizes the fundamental IPT principles into 3-6 sessions. Individuals receiving IPC are initially assessed for symptoms of depression, and then encouraged to identify interpersonal problem areas which may be contributing to their presenting symptoms.
  Other Names: IPC-C

SUMMARY:
Interpersonal Counseling (IPC) is brief, structured modification of Interpersonal Psychotherapy (IPT). IPC was developed as a brief triage manual to treat depression in primary care, family practice and non-mental health programs, and work and educational settings. College and university students are at the age where first episodes of depression, bipolar disorder, or psychosis may occur. IPC is relevant for this population as many university students' distress are related to profound life changes, role transitions, loneliness and social/cultural isolation, which are focuses of treatment in IPC. While there is considerable evidence for the efficacy of IPT and IPC, this adaptation for university students has not yet been studied. The investigators propose to administer IPC to across several college campuses, and to recruit 20 participants at each counseling center. Participants will receive 3-6 one-hour therapy sessions, and will complete self-report measures of depression, psychosocial functioning, college adjustment, and treatment satisfaction. IPC has the potential to reduce depressive symptoms and prevent presenting symptoms from worsening. For these reasons, developing and testing a brief, yet comprehensive psychosocial intervention for distressed college students has tremendous importance.

DETAILED DESCRIPTION:
Interpersonal Psychotherapy (IPT) is a short term, evidence-based treatment approach that has shown benefits in treating major depressive disorder as well as other psychiatric conditions. IPT focuses on the patient's current life events, including social and interpersonal functioning, as a means of understanding and treating maladaptive symptoms. Interpersonal Counseling (IPC) is a modification of the Interpersonal Psychotherapy (IPT) protocol. Subsequently, IPC was developed as a brief intervention for depression to be used in primary care, family practice and non-mental health programs, educational and work settings. IPC is a treatment approach ready for dissemination and implementation by non-mental health workers who have direct contact with individuals at risk for depression and other pathologies. IPC has been used for efficient training, for preventative and screening purposes in doctor's offices, schools, community based centers and organizations.

IPC synthesizes the fundamental principles of IPT into 3-6 sessions. Individuals receiving IPC are initially assessed for symptoms of pathology, and then encouraged to identify interpersonal problem areas which may be contributing to their presenting symptoms. The key principles and techniques standard to IPT are also applied in IPC, so that the protocol can act not only as an assessment tool, but also as a brief intervention. After identifying an interpersonal problem area, the IPC clinician works with the client to mobilize social support and rehearse more effective communication strategies. Once the IPC protocol is completed, clinical decisions can be made regarding clients' need for follow-up psychotherapy or alternative referrals.

Over the last decade, college and university counseling centers are reporting that students are seeking psychiatric services under more distress and with more severe disorders. College-age students are generally at increased risk for experiencing psychopathology; they are at the age where first episodes of depression, bipolar disorder, or psychosis often occur. Secondly, college students are often away from their social and family networks for the first time, and may experience less instrumental social support when experiencing periods of psychological distress. To date, most college counseling centers conduct psychological assessments of students presenting for services and provide supportive counseling, often for a finite number of sessions due to the heavy volume of student referrals. For these reasons, it is important to have a brief, yet comprehensive protocol for screening and intervening with distressed college students. Such protocols should be structured and accessible to implementation by a range of professionals: clinical social workers or psychologists, practicum students and interns training in these fields. IPC, a systematic, brief evaluation, support and triage approach may help university counseling centers in both their treatment and intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Currently receiving counseling at one of the study locations
* Adjustment disorder with depressed mood or mild to moderate depression which correlates with a Patient Health Questionnaire-9 (PHQ-9) score of 5-14.

Exclusion Criteria:

* Pregnancy.
* Non-English speaking
* Poses a significant risk for dangerousness to self or others, or suffers from a concomitant medical or psychiatric comorbidity that makes the study protocol inadvisable (i.e., post-traumatic stress disorder, autism, psychotic disorder, bipolar I or II disorder, eating disorder, alcohol or substance abuse or current use)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Retention rate | One year
  Retention rate will be assessed by calculating the number of participants who completed the study compared to the number of participants who enrolled in the study

SECONDARY OUTCOMES:
Satisfaction questionnaire | Participants complete a satisfaction questionnaire when they have completed the study (maximum of 3 months)
  Assess satisfaction of IPC-C via a 9 question, 7 point likert satisfaction scale questionnaire. High satisfaction with IPC will be evidenced by average scores of 6 on a 7 point satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Miller, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (2):
  - Homewood Counseling Center, Baltimore, Maryland
  - Amherst College Counseling Center, Amherst, Massachusetts
- University of Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No